CLINICAL TRIAL: NCT03709524
Title: A Comparison of Airtraq and Nasotracheal Airtraq for Orotracheal Intubation
Brief Title: Orotracheal Intubation in Adult Patients: A Comparison of Standard Airtraq , Nasotracheal Airtraq Combined With a Stylet Inserted Endotracheal Tube and Standard Airtraq Combined Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KIA 2018/446
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Difficult Intubation
MeSH Terms: interventions — Optical Fibers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insertion time (Active Comparator): 1 minute Airtraq, nasotracheal Airtraq + styletted tube and airtraq + fiberoptic
  Interventions: Device: Airtraq + fiberoptic; Device: Airtraq; Device: Nasotracheal Airtraq + styletted tube
- intubation time (Active Comparator): 2 minutesAirtraq, nasotracheal Airtraq + styletted tube and airtraq + fiberoptic
  Interventions: Device: Airtraq + fiberoptic; Device: Airtraq; Device: Nasotracheal Airtraq + styletted tube

INTERVENTIONS:
Device: Airtraq + fiberoptic — video laryngoscope with a monitor
  Other Names: videolaryngoscope
Device: Airtraq — video laryngoscope with a monitor
  Other Names: videolaryngoscope
Device: Nasotracheal Airtraq + styletted tube — video laryngoscope with a monitor
  Other Names: videolaryngoscope

SUMMARY:
Adult patients requiring endotracheal intubation divided into three groups; standard Airtraq, Nasotracheal Airtraq + styletted endotracheal tube and Airtraq + fiberoptic combination groups.

DETAILED DESCRIPTION:
We enroll lean adult patients requiring endotracheal intubation. Using a sealed envelope technique they divided into three groups; Standard Airtraq and Nasotracheal Airtraq + styletted endotracheal tube and Standard Airtraq + fiberoptic combination. Demographic characteristics and airway management variables such; age, gender, height, weight, ASA status, tooth morphology, tiro mental and sternomental distance were recorded. Insertion times, intubation times and total intubation times with these devices will be recorded. Hemodynamic parameters recorded such as; heart rate will be recorded baseline , after anesthesia, after insertion, just after and then every 2 minutes intervals after intubation. sore throat, hoarseness, dysphasia, bronchospasm were also recorded postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* BMI<30
* > 18 AGE
* requiring endotracheal intubation
* ASA 1-2

Exclusion Criteria:

* BMI> 30
* < 18 AGE
* ASA III-IV
* upper respiratory infection past ten days
* pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Intubation time | 6 months
  entering the oral cavity till intubation

SECONDARY OUTCOMES:
insertion time | 6 months
  entering the oral cavity till the optimal visualization

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No